CLINICAL TRIAL: NCT01708876
Title: Artesunate-mefloquine vs Chloroquine in Patients With Acute Uncomplicated P. Knowlesi and P. Vivax Malaria: a Randomized Open Label Trial in Sabah, Malaysia
Brief Title: P. Knowlesi Trial of Artesunate-mefloquine Versus Chloroquine
Acronym: ACT KNOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-12-89-11005
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Uncomplicated Plasmodium Knowlesi Malaria
Keywords: uncomplicated; plasmodium; knowlesi; malaria; infection
MeSH Terms: conditions — Malaria; Infections | interventions — Chloroquine; Alkalies; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artesunate-mefloquine (Active Comparator): 3 doses artesunate-mefloquine - daily over 3 days (dosage according to bodyweight - 4mg/kg and 8.3mg/kg respectively).
  Interventions: Drug: Artesunate-mefloquine; Drug: Primaquine
- Chloroquine (Active Comparator): 4 doses chloroquine over 3 days - total dose 25mg/kg. 10mg/kg at 0 hours, 5mg/kg at 6-8, 24, 48 hours.
  Interventions: Drug: Chloroquine; Drug: Primaquine

INTERVENTIONS:
Drug: Artesunate-mefloquine
  Other Names: Artequin 600/1500; Artequin 300/750; Artequin Paed granules 50/125
  Arms: Artesunate-mefloquine
Drug: Chloroquine
  Other Names: Chloroquine; 1 tablet = 155mg base
  Arms: Chloroquine
Drug: Primaquine — Given to P. vivax patients only. Delayed administration at day 28; 0.5mg/kg for children or 45mg for adults; normal G6PD activity (once daily administration for 14 days); moderate G6PD deficiency (once weekly for 8 weeks); severe G6PD deficiency (contraindicated / not given).

SUMMARY:
Preliminary studies have supported the background efficacy of local standard anti-malarial medications in the treatment of uncomplicated knowlesi malaria, however this has not been tested systematically and there are no current WHO treatment guidelines for this infection. There are both health cost benefits to a more rapidly acting agent, and due to difficulties with microscopic identification there may be more effective treatment for all malaria species if an aligned treatment guideline could be supported. In addition, no therapeutic efficacy monitoring of current first line anti-malarials used for the treatment of P. vivax malaria have been conducted in Malaysia.

The investigators aim to test whether the fixed combination of artesunate-mefloquine is superior to chloroquine in order to define the optimal treatment for both uncomplicated P. knowlesi and P. vivax infection in both adults and children in this region.

DETAILED DESCRIPTION:
1.1 Background

Naturally acquired infections with Plasmodium knowlesi, the fifth human malaria, are growing [1]. Since 2004 increasing numbers of cases have been reported from residents and returned travelers predominantly from Malaysia and other countries in South-East Asia including Thailand, Vietnam, Myanmar, Singapore, Indonesia and the Philippines [2-8]. Cases coincide with the geographic distribution of its natural simian hosts (long-tailed and pig-tailed macaques) and Anopheles leucosphyrus group mosquito vector [9, 10], with potential human-to-human transmission unknown. Eastern Malaysia appears to be the epicentre, with around 1400 PCR-confirmed P. knowlesi human mono-infections reported in 2009, comprising 41% of 2,189 total malaria cases in Sarawak [11] and 343 cases from selected samples sent to Sabah's State Reference Laboratory [12]. P. knowlesi is also now the most common cause of malaria in different contrasting regions, including 70% of malaria admissions in the heavily forested area of Kapit in Sarawak [1, 13], 63% of samples from the interior division of Sabah [14], and in 87% of malaria admissions in the deforested coastal area of Kudat in Sabah, where it is also the major cause of malaria in children [15].

Despite the increase in reported incidence, difficulties with microscopic diagnosis and a lack of PCR based epidemiological surveillance studies throughout South-East Asia mean the true disease burden is underestimated. P. knowlesi is microscopically misidentified as P . falciparum and P. malariae due to morphological similarities in the early trophozoite, and late trophozoite and schizont life stages respectively, with studies showing up to 80% of P. malariae [16-19] and 7-12% of P. falciparum [1, 16] in this region are actually P. knowlesi when definitively evaluated with PCR. Current rapid diagnostic tests (RDT) for malaria can distinguish falciparum Current rapid diagnostic tests (RDT) for malaria can distinguish falciparum from other Plasmodium species with a sensitivity of up to 99% at parasite counts > 1,000/ μL [20], but a knowlesi specific antigen has not been developed and current antibody panels are unable to differentiate between P. knowlesi and other mixed Plasmodium spp. infections [21]. Misdiagnosis has concerning treatment implications, as unlike P. malariae, knowlesi malaria has a rapid 24-hour replication rate and can cause hyperparasitaemia, severe complications and fatal outcomes [13, 17, 18], while the inadvertent use of chloroquine for widely chloroquine-resistant P. falciparum may also have fatal consequences.

1.2 Treatment

Initial observational and retrospective studies have suggested both chloroquine and artemisinin combination therapy (ACT) are effective therapy for uncomplicated P. knowlesi infection [15, 16, 22, 23]. Justification for treatment selection for this trial is based on this literature review. Case reports predominantly from returned travelers to South-East Asia also document uncomplicated knowlesi malaria responding well to conventional anti-malarials such as chloroquine, mefloquine, atovaquone with proguanil, doxycycline and quinine [4, 24- 31], supporting its zoonotic and drug naïve origin. However to date there have been no prospective randomised trials to compare chloroquine and ACT as the anti-malarials currently used for uncomplicated P. knowlesi infection in Malaysia, and there are no current recommendations on how to treat P. knowlesi infection in the WHO 2010 malaria treatment guidelines. As ACTs are already being used for treating P. falciparum and are recommended for the increasingly chloroquine-resistant P. vivax found in the surrounding countries in South East Asia [32], the potential benefit of a unified treatment policy to facilitate prompt and effective treatment of all Plasmodium species needs evidence of ACT as the optimal treatment for P. knowlesi infection also.

Malaysian Ministry of Health guidelines currently recommend chloroquine and primaquine as first line treatment for the erythrocytic and hypnozoite life stages of uncomplicated P. vivax malaria respectively. While resistance to chloroquine has previously been documented in Sabah [35] and Peninsular Malaysia [36-38], the unstable transmission dynamics and recent reduction in P. vivax incidence due to public health measures mean the current risk of chloroquine-resistant P.vivax transmission is likely to be low. Despite this, due to increasing resistance in surrounding countries including Indonesia, Thailand, Vietnam, and PNG [39], transient populations of migrant workers, and recent concerns of the failing efficacy of hypnozoite eradication by primaquine [40], the need for ongoing therapeutic efficacy monitoring is recommended [41].

1.3 Artesunate-mefloquine

Artesunate-mefloquine (AS-MQ) is a common and widely available ACT, and along with artemether-lumefantrine (A-L) is one of only 2 first line WHO recommended options for the treatment of uncomplicated P. falciparum infection which are registered in Malaysia and produced according to international good manufacturing practice (GMP) standards. ACTs are the current mainstay of malaria elimination efforts [33], with a mechanism of action resulting both in a rapid reduction in parasite mass and resolution of clinical features, while the long acting component eliminates residual parasites and delays the development of de novo resistance [34, 35]. Safety and tolerability of all ACTs are dependent on their partner drug [36], and while gastro-intestinal and self-limiting neuro-psychiatric adverse events have been reported with mefloquine, multiple safety and efficacy trials have recommended its use in both adults and children for uncomplicated falciparum malaria [37-40]. Due to concerns over the safety of mefloquine in the first trimester of pregnancy [41], and its use in patients with pre-existing psychiatric disorders or those who have previously had cerebral malaria, it is currently not advised for these groups [36].

The only reported use of ACT for knowlesi malaria is from our retrospective study at a tertiary referral hospital in Sabah, where a small sample size of 8 out of 34 patients with PCR- confirmed uncomplicated P. knowlesi infection were treated with oral artemether- lumefantrine. Median microscopic parasite clearance time was 1 day (range 0-3), which was significantly faster than those receiving chloroquine (median 2.5 days, range 1-3, p = 0.01) [23]. There are no published reports of other ACTs used in the treatment of P. knowlesi infection, although currently both AS-MQ and A-L are being used in Sabah for uncomplicated P. knowlesi and P. falciparum malaria, including in children >5kg, as recommended by local guidelines.

Mefloquine as a single agent has also been used in the successful treatment of a Swedish traveller returning from Sarawak, Malaysia with PCR confirmed uncomplicated P. knowlesi infection in 2009 [24]. The long half life of mefloquine of around 14 days also means when used as the partner drug in an ACT for uncomplicated malaria caused by other Plasmodium species such as P. vivax, there is a significant reduction compared to A-L in the day 42 treatment failure rate [42].

1.4 Chloroquine

Chloroquine with primaquine was initially suggested to have favourable treatment outcomes for uncomplicated P. knowlesi human infections after a retrospective review of patients from Kapit Hospital in Sarawak in 2004 [16]. Following this a single prospective observational study conducted at the same site between 2006-7 administered chloroquine as a total base dose of 25mg/kg and primaquine as a gametocidal agent to 73 patients with uncomplicated PCR-confirmed P. knowlesi malaria, with results showing median fever clearance of 26 hours, mean times to 50% and 90% microscopic parasite clearance of 3.1 and 10.3 hours respectively, and a median PCR adjusted clearance time of 3 days. None of the 60 patients who completed the 28-day follow up demonstrated any evidence of resistance, re-infection or recrudescence [22].

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 1 year of age and weighing more than 10kg
* Microscopic diagnosis of Plasmodium species infection
* Negative P. falciparum malaria rapid diagnostic test (histidine rich protein 2)
* Fever (temperature 37.5°C) or history of fever in the last 48 hours
* Able to participate in the trial and comply with the clinical trial protocol
* Written informed consent to participate in trial; thumbprint is required for illiterate patients, and written consent from parents/guardian for children below age of consent

Exclusion Criteria:

* Clinical or laboratory criteria for severe malaria, including warning signs, requiring parenteral treatment according to modified WHO criteria (see Appendix 4)
* Parasitaemia > 20,000 /μL (P. knowlesi)
* Inability to tolerate oral treatment
* Concomitant infection with any other malaria species
* Pregnancy or lactation
* Unable or unwilling to use contraception during study period
* Known hypersensitivity or allergy to artemisinin derivatives
* Serious underlying disease (cardiac, renal or hepatic)
* Received anti-malarials in last 2 months
* Previous psychiatric illness or epilepsy
* Previous episode of cerebral malaria

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Parasite clearance | 24 hours
  The primary endpoint is the therapeutic efficacy of artesunate-mefloquine versus chloroquine, as defined by the assessment of microscopic P. knowlesi and P. vivax parasite clearance 24 hours after initiation of treatment.

SECONDARY OUTCOMES:
Rates of recurrent infection / treatment failure at day 42. | 42 days
Occurrence of anaemia at day 28 when using AS-MQ vs. CQ. | 28 days
P. knowlesi and P. vivax gametocyte carriage throughout follow up when using AS-MQ vs. CQ. | 42 days
Frequency of complications throughout follow up when using AS-MQ vs. CQ. | 42 days
Utility of malaria rapid diagnostic tests in diagnosis of P. knowlesi infection. | 1 day
Rates of P. knowlesi and P. vivax recurrence in a 1 year follow up period. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jayaram Menon, MBBS, Study Director — Sabah Ministry of Health; D Prabhakaran, MBBS, Study Director — Sabah Ministry of Health; Matthew J Grigg, MBBS, Study Director — Menzies School of Health Research; Tsin Yeo, MBBS, Study Director — Menzies School of Health Research; Lorenz von Seidlein, MBBS, Study Director — Menzies School of Health Research; Nicholas M Anstey, MBBS, Study Director — Menzies School of Health Research; Ric Price, MBBS, Study Director — Menzies School of Health Research
Locations (3):
- Malaysia (3):
  - Kota Marudu District Hospital, Kota Marudu, Sabah
  - Kudat District Hospital, Kudat, Sabah
  - Pitas District Hospital, Pitas, Sabah

REFERENCES:
- [Background] Putaporntip C, Hongsrimuang T, Seethamchai S, Kobasa T, Limkittikul K, Cui L, Jongwutiwes S. Differential prevalence of Plasmodium infections and cryptic Plasmodium knowlesi malaria in humans in Thailand. J Infect Dis. 2009 Apr 15;199(8):1143-50. doi: 10.1086/597414. PMID 19284284
- [Background] Marchand RP, Culleton R, Maeno Y, Quang NT, Nakazawa S. Co-infections of Plasmodium knowlesi, P. falciparum, and P. vivax among Humans and Anopheles dirus Mosquitoes, Southern Vietnam. Emerg Infect Dis. 2011 Jul;17(7):1232-9. doi: 10.3201/eid1707.101551. PMID 21762577
- [Background] Ng OT, Ooi EE, Lee CC, Lee PJ, Ng LC, Pei SW, Tu TM, Loh JP, Leo YS. Naturally acquired human Plasmodium knowlesi infection, Singapore. Emerg Infect Dis. 2008 May;14(5):814-6. doi: 10.3201/eid1405.070863. PMID 18439370
- [Background] Jiang N, Chang Q, Sun X, Lu H, Yin J, Zhang Z, Wahlgren M, Chen Q. Co-infections with Plasmodium knowlesi and other malaria parasites, Myanmar. Emerg Infect Dis. 2010 Sep;16(9):1476-8. doi: 10.3201/eid1609.100339. PMID 20735938
- [Background] Vythilingam I. Plasmodium knowlesi in humans: a review on the role of its vectors in Malaysia. Trop Biomed. 2010 Apr;27(1):1-12. PMID 20562807
- [Background] Figtree M, Lee R, Bain L, Kennedy T, Mackertich S, Urban M, Cheng Q, Hudson BJ. Plasmodium knowlesi in human, Indonesian Borneo. Emerg Infect Dis. 2010 Apr;16(4):672-4. doi: 10.3201/eid1604.091624. PMID 20350383
- [Background] Luchavez J, Espino F, Curameng P, Espina R, Bell D, Chiodini P, Nolder D, Sutherland C, Lee KS, Singh B. Human Infections with Plasmodium knowlesi, the Philippines. Emerg Infect Dis. 2008 May;14(5):811-3. doi: 10.3201/eid1405.071407. PMID 18439369
- [Background] Baird JK. Malaria zoonoses. Travel Med Infect Dis. 2009 Sep;7(5):269-77. doi: 10.1016/j.tmaid.2009.06.004. Epub 2009 Jul 14. PMID 19747661
- [Background] Singh B, Daneshvar C. Plasmodium knowlesi malaria in Malaysia. Med J Malaysia. 2010 Sep;65(3):166-72. PMID 21939162
- [Result] Cox-Singh J, Davis TM, Lee KS, Shamsul SS, Matusop A, Ratnam S, Rahman HA, Conway DJ, Singh B. Plasmodium knowlesi malaria in humans is widely distributed and potentially life threatening. Clin Infect Dis. 2008 Jan 15;46(2):165-71. doi: 10.1086/524888. PMID 18171245
- [Derived] Longley RJ, Grigg MJ, Schoffer K, Obadia T, Hyslop S, Piera KA, Nekkab N, Mazhari R, Takashima E, Tsuboi T, Harbers M, Tetteh K, Drakeley C, Chitnis CE, Healer J, Tham WH, Sattabongkot J, White MT, Cooper DJ, Rajahram GS, Barber BE, William T, Anstey NM, Mueller I. Plasmodium vivax malaria serological exposure markers: Assessing the degree and implications of cross-reactivity with P. knowlesi. Cell Rep Med. 2022 Jun 21;3(6):100662. doi: 10.1016/j.xcrm.2022.100662. PMID 35732155
- [Derived] Grigg MJ, William T, Menon J, Barber BE, Wilkes CS, Rajahram GS, Edstein MD, Auburn S, Price RN, Yeo TW, Anstey NM. Efficacy of Artesunate-mefloquine for Chloroquine-resistant Plasmodium vivax Malaria in Malaysia: An Open-label, Randomized, Controlled Trial. Clin Infect Dis. 2016 Jun 1;62(11):1403-1411. doi: 10.1093/cid/ciw121. Epub 2016 Apr 22. PMID 27107287
- [Derived] Grigg MJ, William T, Menon J, Dhanaraj P, Barber BE, Wilkes CS, von Seidlein L, Rajahram GS, Pasay C, McCarthy JS, Price RN, Anstey NM, Yeo TW. Artesunate-mefloquine versus chloroquine for treatment of uncomplicated Plasmodium knowlesi malaria in Malaysia (ACT KNOW): an open-label, randomised controlled trial. Lancet Infect Dis. 2016 Feb;16(2):180-188. doi: 10.1016/S1473-3099(15)00415-6. Epub 2015 Nov 19. PMID 26603174
- [Derived] Grigg MJ, William T, Dhanaraj P, Menon J, Barber BE, von Seidlein L, Rajahram G, Price RN, Anstey NM, Yeo TW. A study protocol for a randomised open-label clinical trial of artesunate-mefloquine versus chloroquine in patients with non-severe Plasmodium knowlesi malaria in Sabah, Malaysia (ACT KNOW trial). BMJ Open. 2014 Aug 19;4(8):e006005. doi: 10.1136/bmjopen-2014-006005. PMID 25138814